CLINICAL TRIAL: NCT06105788
Title: Comparing Effects of Upper Extremity Versus Lower Extremity Exercise on Exercise-Induced Hypoalgesia in People With Knee Osteoarthritis: A Pilot Cross-over Study
Brief Title: Upper and Lower Extremity Exercise and Exercise-Induced Hypoalgesia in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2111266
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Central Pain Syndrome
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise; Exercise Test

STUDY DESIGN:
Intervention Model Description: This will be a pilot randomized cross-over study. Once enrolled, all participants will undergo 3 laboratory visits, each separated at least by a week as a wash-out period: day 1, baseline assessment; day 2, randomized to either arm exercise (AE) or leg exercise (LE) ; and day 3, AE or LE alternative to the exercise on day 2.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Arm 1: All participants, knee OA and pain-free individuals, will undergo a single exercise of arm exercise using an arm ergometer and;
  Interventions: Other: Exercise
- Lower Body Exercise (Active Comparator): Arm 2: All participants, knee OA and pain-free individuals, will undergo a single exercise of leg exercise using a cycling ergometer.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Arm exercise will be an arm ergometer for 20 minutes, preceded by a 5-minute warm-up.
  Leg exercise will be a cycling ergometer for 20 minutes, preceded by a 5-minute warm-up.
  The exercise intensity will be set at 70% of the heart rate reserve (HRR) for each type of exercise.
  Other Names: Arm exercise; Leg exercise

SUMMARY:
The objective of the study is to explore the effects of arm exercise (UE, arm ergometer) vs. leg exercise (LE, cycling ergometer) on exercise-induced hypoalgesia (EIH), central pain mechanisms and knee pain in people with knee osteoarthritis (OA). Furthermore, we will explore relations of socioeconomic status, racial discrimination, acculturative stress, and autonomic function to exercise effects on EIH, central pain mechanisms, and knee pain. This will be a pilot randomized cross-over study where all participants undergo Day 1 (baseline assessments), Day 2 (UE or LE), and Day 3 (UE or LE).

DETAILED DESCRIPTION:
This will be a pilot randomized cross-over study. Major exclusion criteria will be conditions that have risks with exercise or affect pain assessments. Once enrolled, all participants will undergo 3 laboratory visits, each separated at least by a week as a wash-out period: day 1, baseline assessment; day 2, randomized to either upper extremity exercise (UEE) (i.e., arm ergometer) or knee exercise (KE) (i.e., cycling ergometer); and day 3, UEE or KE alternative to the exercise on day 2. UEE will be an arm-ergometer and KE will be a cycle-ergometer in which participants will undergo the first 5 minutes at an intensity of 50% heart rate reserve (HRR)(warm-up period), followed by 20 minutes at 70% HRR. Heart rate will be monitored during the exercise.

On day 1, we will collect participant characteristics data. We will also collect data related to race/ethnicity, racial discrimination, acculturative stress, physical activity level, heart rate variability (HRV) parameters (measures of autonomic function). Further, participants will undergo knee pain assessment with a 20-meter walk, quantitative sensory testing (QST) measures of pressure pain threshold (PPT), temporal summation (TS), and conditioned pain modulation (CPM) as surrogate measures of central pain mechanisms.

On Days 2 and 3 we will collect knee pain, QST, and EIH data before and immediately after the exercise.

ELIGIBILITY:
Participants with knee OA (Target n=40)

Inclusion Criteria:

We will recruit participants with knee OA, using the National Institute for Health and Care Excellence's clinical diagnostic criteria, which does not require radiographs. The clinical diagnostic criteria include:

* age ≥45
* activity-related knee pain
* either no morning joint-related stiffness or stiffness that lasts ≤ 30 minutes.
* knee pain at least 4 on a 0-10 pain scale
* knee pain as a chief complaint if having multiple pain
* understand English

Exclusion Criteria:

* peripheral neuropathy or other sensation loss on the body sites for pain measurements (i.e., the wrist, knee, the forearm)
* use of medical devices electrically active (e.g., pacemaker)
* chronic use of opioids
* pregnant women
* serious and uncontrolled concomitant disease, including cardiovascular, nervous system, pulmonary, renal, hepatic, metabolic, hormonal, endocrine, gastrointestinal or epileptic disease
* rheumatoid arthritis, ankylosing spondylitis, and any neurological disorders that prevent the study procedure
* cognitive impairment
* history of a knee replacement surgery
* inability to perform exercise due to severe pain or other symptoms
* any intervention procedures for knee pain in the last 3 months

Inclusion and exclusion criteria for pain-free controls (Target n = 20) Pain-free controls are not having a pain-related medical condition. They have to speak and understand English. Pain-free controls are excluded if they had experienced a pain episode, caused by musculoskeletal injury or otherwise in the previous 3 months.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-10-16 (Estimated)

PRIMARY OUTCOMES:
Changes in pressure pain thresholds (Measure of exercise-induced hypoalgesia) | Day 1: PPT will be assessed twice. PPT assessment --> 25 minutes of waiting --> PPT assessment; Time frame of Days 2 and 3 will be the same except 25 minutes of waiting time. It will be 25 minutes of exercise (either AE or LE) on Days 2 and 3
  Pressure pain thresholds (PPT) will be assessed at the wrist and patella. PPT being assessed at a remote body site (e.g., wrist) is to measure central pain sensitivity while PPT being assessed at the location of pain (i.e., knee, patellae) is to assess peripheral pain sensitivity with or without central pain sensitivity. PPT will be assessed using a handheld pressure algometer with 1 cm2 rubber tip. PPT will be defined as the point at which the participant verbally indicated that the pressure first changed to slight pain. A lower PPT value (Kgf) represents greater pain sensitivity. PPT will be assessed 3 times at each location and averaged. Furthermore, changes in PPT after exercise has been used to assess the degree of exercise-induced hypoalgesia (EIH). When PPT values increase after the exercise, it indicates a reduction of pain sensitivity and, therefore, an effect of EIH.
Mechanical temporal summation | Day 1: TS will be assessed twice. TS assessment --> 25 minutes of waiting --> TS assessment; Time frame of Days 2 and 3 will be the same except 25 minutes of waiting time. It will be 25 minutes of exercise (either AE or LE) on Days 2 and 3
  Temporal summation (TS) is a sensitive measurement of central pain sensitivity. Investigators will assess TS using a standard set of weighted probes from 64-512 mN. Participants will rate the pain experienced by each successive weighted probe being touched on the skin of the wrist until a pain rating of ≥ 4/10 is achieved. The selected probe will be then applied at a frequency of 1 Hz for 10 seconds on the wrist. Participants will provide a pain rating at the completion of the train of 10 stimulations and 15 seconds post-stimulation. TS will be defined as the difference between the highest post-stimulation pain rating and the initial pain rating. A post-stimulation pain rating greater than the initial pain rating will be considered to be reflective of an increase in central pain sensitivity.
Conditioned pain modulation | Day 1: CPM will be assessed twice. CPM assessment --> 25 minutes of waiting --> CPM assessment; Time frame of Days 2 and 3 will be the same except 25 minutes of waiting time. It will be 25 minutes of exercise (either AE or LE) on Days 2 and 3
  Conditioned pain modulation (CPM) evaluates the adequacy of the descending pain modulatory pathways, which contributes to central pain sensitivity. Investigators will assess CPM using PPT as the test stimulus (PPT1) at the wrist as described above, with forearm ischemia using a blood pressure cuff as the conditioning stimulus. Briefly, the blood pressure cuff applied to the contralateral arm will be inflated to 10mm Hg above systolic pressure. The participant will be then instructed to perform hand grip squeezes until pain of at least 4/10 occurs in the contralateral arm. PPT will be then reassessed at the wrist 3 times and averaged (PPT2). Percent efficiency of CPM (%CPM) was computed as PPT2/PPT1, multiplied by 100; %CPM ≤ 100 indicates inefficient CPM.
Knee pain | Day 1: knee pain will be assessed twice. Knee pain assessment --> 25 minutes of waiting --> knee pain assessment; Time frame of Days 2 and 3 will be the same except 25 minutes of waiting time. It will be 25 minutes of exercise (either AE or LE) on Days 2
  We will assess changes in knee pain with a 20 meter walk using a 0-10 numeric rating scale where 0 indicates no knee pain and 10 indicates the worst knee pain.

SECONDARY OUTCOMES:
Racial discrimination | Day 1 after obtaining the informed consent form
  Racial discrimination will be assessed with the Perceived Experiences of Discrimination Questionnaire-Community Version (PEDQ-CV). This is a reliable and valid 17-item survey that assesses experiences of racialized discrimination.
Acculturative Stress | Day 1 after obtaining the informed consent form
  Acculturative stress will be assessed with The Social, Attitudinal, Familial, Environment Acculturative Stress Scale (SAFE). SAFE is composed of 24 items that measure stress as a result of the acculturation process in four contexts: social, attitudinal, familial and environmental acculturative.
Autonomic function | Day 1 after obtaining the informed consent form
  Heart rate variability (HRV), a measurement of autonomic function, will be assessed using a wearable and wireless heart rate monitor. Investigators will have participants lie supine for 5 minutes to collect heart rate variability parameters such as high frequency and high-frequency/low-frequency ratio.
The Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) | Day 1 after obtaining the informed consent form
  WOMAC knee pain scale ranges 0-20 with 5 questions assessing knee pain in different contexts such as knee pain during walking and pain during standing. Each question has a score of 0-4. A greater WOMAC score represents greater knee pain.
Pain catastrophizing scale (PCS) | Day 1 after obtaining the informed consent form
  The Pain Catastrophizing Scale is a validated 13-item scale with questions related to catastrophizing behavior. The total score is 52 with higher scores indicating greater catastrophic thoughts.
Pittsburgh sleep quality index (PSQI) | Day 1 after obtaining the informed consent form
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire. PSQI contains 19 individual items, creating seven components that produce one global score, ranging from 0 to 21. A score of 0-4 indicates the absence of sleep problems, while scores 5 and higher indicate poor sleep quality.
Hospital anxiety and depression scale (HADS) | Day 1 after obtaining the informed consent form
  HADS contains seven questions about anxiety and seven questions about depression, with a 0-3 score for each question. Higher scores indicate greater anxiety and depression.
Physical activity | Day 1 after obtaining the informed consent form
  Physical activity will be assessed with International Physical Activity Questionnaire (IPAQ). IPAQ is a 27-item self-reported measure of physical activity. Results can be reported in categorical (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Instrument support | Day 1 after obtaining the informed consent form
  Instrument support will be assessed with the PROMIS SFv2.0 Instrumental Support 6a questionnaire. This is a 6-item questionnaire with a 5-point Likert scale ranging from "never" to "Always". Each score will be standardized to T-scores with mean of 50 standard deviation of 10. A higher score indicates having more support.
Emotional support | Day 1 after obtaining the informed consent form
  Emotional support will be assessed with the PROMIS SFv2.0 Emotional Support 6a questionnaire. This is a 6-item questionnaire with a 5-point Likert scale ranging from "never" to "Always". Each score will be standardized to T-scores with mean of 50 standard deviation of 10. A higher score indicates having more support.
Positive and negative affect | Day 1 after obtaining the informed consent form
  The Positive and Negative Affect Schedule (PANAS) is a 20-item measure that consists of 10 positive items (e.g., excited, proud) and 10 negative items (e.g., distressed, scared). Items are self-rated on a 5-point Likert-type scale ranging from 1 (very slightly or not at all) to 5 (extremely) and summed to produce total subscale scores for positive and negative affect ranging from 10 to 50, with higher scores representing higher levels of each subscale

CONTACTS AND LOCATIONS:
Overall Officials: Kosaku Aoyagi, PhD, Principal Investigator — Assistant Professor
Locations (1):
- The University of Texas at El Paso, El Paso, Texas, United States